CLINICAL TRIAL: NCT00002179
Title: A Multiclinic, Open Study to Evaluate the Ability of the Combination of Indinavir, Zidovudine and Lamivudine to Result in Sustained Suppression of HIV-1 in Asymptomatic HIV-1 Seropositive Patients
Brief Title: The Effectiveness of Indinavir Plus Zidovudine Plus Lamivudine in HIV-Infected Patients With No Symptoms of Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246G; MK-0639
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Semen; Monocytes; HIV-1; Drug Therapy, Combination; Zidovudine; Lymph Nodes; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To evaluate the ability of the combination of indinavir, zidovudine, and lamivudine to suppress HIV-1 infection as measured by: (1) the maintenance of HIV-1 serum viral RNA below the limit of detection of the most sensitive validated assay (ultradirect assay) and (2) absence of evidence of infectious virus in lymph node, cerebrospinal fluid (CSF), peripheral mononuclear cells (PBMCs), and semen.

It is hypothesized that the administration of indinavir, zidovudine, and lamivudine will result in:

1. No evidence of infectious virus in lymph node tissue, CSF, PBMCs, and semen samples in 50% of patients who have undetectable viral RNA by the most sensitive validated assay available (ultradirect assay) for at least 48 weeks.
2. Sustained suppression of HIV-1 infection as measured by a decrease in serum viral RNA to below the limit of detection of the ultradirect assay for at least 48 weeks in at least 25% of patients.
3. Suppression of HIV-1 infection as measured by a decrease in serum viral RNA to below the limit of detection of the standard Amplicor assay (i.e., negative) in at least 90% of patients by Week 16.
4. Suppression of HIV-1 infection, suggesting eradication of the virus as measured by maintenance of serum viral RNA to below the limit of detection of the ultradirect assay for at least 24 weeks after discontinuation of indinavir, zidovudine, and lamivudine in patients who have maintained this level of suppression for at least 120 weeks on therapy.

DETAILED DESCRIPTION:
It is hypothesized that the administration of indinavir, zidovudine, and lamivudine will result in:

1. No evidence of infectious virus in lymph node tissue, CSF, PBMCs, and semen samples in 50% of patients who have undetectable viral RNA by the most sensitive validated assay available (ultradirect assay) for at least 48 weeks.
2. Sustained suppression of HIV-1 infection as measured by a decrease in serum viral RNA to below the limit of detection of the ultradirect assay for at least 48 weeks in at least 25% of patients.
3. Suppression of HIV-1 infection as measured by a decrease in serum viral RNA to below the limit of detection of the standard Amplicor assay (i.e., negative) in at least 90% of patients by Week 16.
4. Suppression of HIV-1 infection, suggesting eradication of the virus as measured by maintenance of serum viral RNA to below the limit of detection of the ultradirect assay for at least 24 weeks after discontinuation of indinavir, zidovudine, and lamivudine in patients who have maintained this level of suppression for at least 120 weeks on therapy.

All patients receive indinavir plus zidovudine plus lamivudine for at least 96 weeks. If there is no evidence of infectious virus, and patients continue to have serum viral RNA levels below the limit of detection of the ultradirect assay for at least 96 weeks, therapy is continued for an additional 24 weeks. However, during this additional 24 weeks of therapy patients may continue to receive this triple combination drug regimen or make changes to this drug regimen treatment by reducing their number of antiretroviral agents. After 120 weeks, if patients continue to have serum viral RNA levels below the limit of detection of the ultradirect assay, patients discontinue all antiretroviral therapy. However, if there is any evidence of infectious virus, as outlined above, patients do not discontinue therapy. Patients who develop detectable serum viral RNA following discontinuation of therapy are given the option to reinitiate therapy with the triple combination of indinavir, zidovudine and lamivudine. NOTE: Patients who develop an intolerance to zidovudine may use stavudine at doses per body weight at the direction of the investigator.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositive status.
* CD4 count >= 500 cells/mm3.
* Serum viral RNA level > 1000 copies/ml.

Exclusion Criteria

Prior Medication:

Excluded:

Previous antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - LAC - USC Med Ctr, Los Angeles, California
  - AIDS Community Research Consortium, Redwood City, California
  - San Francisco Gen Hosp, San Francisco, California
  - Yale Univ School of Medicine / AIDS Program, New Haven, Connecticut
  - Rush Presbyterian - Saint Luke's Med Ctr / Infect Dis, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Fenway Community Health Ctr, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr - East Campus, Boston, Massachusetts
  - NYU Med Ctr, New York, New York
  - Univ Hosp / SUNY at Stony Brook / AIDS TMT Unit, Stony Brook, New York
  - Pitt Treatment Ctr, Pittsburgh, Pennsylvania
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
- Canada (2):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Montreal Gen Hosp, Montreal, Quebec